CLINICAL TRIAL: NCT00814606
Title: A Pilot Trial to Determine the Safety and Efficacy of Fluvastatin in Previous Partial Responders to Pegylated Interferon and Ribivirin in Patients With Genotype 1 Hepatitis C
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no one ever enrolled
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16336A
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis C; Hepatitis C Virus
Keywords: genotype 1 hepatitis C; hepatitis C; HCV; liver
MeSH Terms: conditions — Hepatitis C | interventions — Fluvastatin; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group (Experimental): 8 weeks period of escalating doses of fluvastatin to a goal dose of 80mg daily, then patients will start treatment of HCV at week 9 with the usual standard of care protocol for medication dose, office visits and laboratories. Peginterferon alfa2a 180 mcg/ml SQ injection once a week for 48 weeks and ribavirin 1000-1200 mg daily orally in two divided doses for 48 weeks. Patients weighing < 75 kg will receive 1000mg per day (400mg in the morning and 600mg in the evening). Patients weighing ≥ 75 kg will receive 1200 mg per day (600mg in the morning and 600 mg in the evening).
  Interventions: Drug: Fluvastatin; Drug: Peginterferon alfa2a; Drug: ribavirin

INTERVENTIONS:
Drug: Fluvastatin — Week 1: Fluvastatin 20mg daily Week 3: Fluvastatin 40mg daily Week 5: Fluvastatin 60mg daily Week 7: Fluvastatin 80 mg daily
Drug: Peginterferon alfa2a — 180 mcg/ml SQ injection once a week for 48 weeks (starting at week 9)
  Other Names: Pegasys
Drug: ribavirin — 1000-1200 mg daily orally in two divided doses for 48 weeks (starting at week 9)
  Other Names: Copegus

SUMMARY:
This study seeks to evaluate the safety and efficacy of taking fluvastatin along with peginterferon alfa in previous partial responders with genotype 1 HCV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any ethnicity age 18 - 65 years with genotype 1 HCV
* Previous partial responder to attempts at HCV therapy with PEG/RBV (at least 1 log drop but less than 2 log drop in HCV RNA at 12 weeks)
* Previous history or serum HCV-RNA PCR quantifiable by Roche Amplicore HCV Test
* A liver biopsy within 3 years of study enrollment consistent with HCV disease.
* Compensated liver disease, Child-Pugh Class ≤ 6
* Negative urine pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of the study drug
* All patients enrolling in the study and all partners of study participants of childbearing potential must be using two reliable forms of effective contraception during the study. Exceptions may include partner/participant is surgically sterile.
* Willingness to comply with study procedures and provide written informed consent

Exclusion Criteria:

* AST or ALT > 10 ULN
* Any investigational drug ≤ 12 weeks prior to the first of study drug
* Prior intolerance to statin medications
* Previous serious side effects to IFN or RBV (e.g. psychiatric side effect necessitating treatment discontinuation, severe cytopenia refractory to growth factors, intolerance to IFN/RBV requiring treatment discontinuation)
* Any systemic antiviral therapy ≤ 24 weeks prior to the first dose of study drug or expectation that such treatment will be needed at any time during the study. Exception: Patients who have taken or are expected to require such treatment for herpetic lesions
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc-IgM Ab ,or anti-HIV Ab
* Serum concentrations of cerulplamin or alph-1-antitrypsin consistent with an increased risk of metabolic liver disease
* History or other evidence of a medical condition associated with chronic liver disease (e.g. hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure, nonalcoholic steatohepatitis)
* Women who are pregnant or breastfeeding and male partners of woman who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of adding fluvastatin to pegylated interferon alfa-2a and ribavirin in patients infected with genotype 1 HCV who are previous partial responders to standard treatment. | 18 months

SECONDARY OUTCOMES:
Safety of adding fluvastatin to pegylated interferon alfa-2a and ribavirin in patients infected with genotype 1 HCV who are previous partial responders to standard treatment. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: K Gautham Reddy, MD, Principal Investigator — University of Chicago